CLINICAL TRIAL: NCT06458725
Title: Comprehensive Assessment of Diffusion-Weighted Magnetic Resonance Imaging (DW-MRI) Measures: Reproducibility and Repeatability in Pelvic Imaging on MR-Linac With Healthy Volunteers. (PILLAR)
Brief Title: Assessment of DW-MRI Measures : Reproducibility and Repeatability in Pelvic Imaging on MR-Linac With Healthy Volunteers
Acronym: PILLAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B0792024000002
Record Dates: First submitted 2024-05-08; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-04

CONDITIONS: Rectum Cancer; Pelvic Cancer
Keywords: Repeatability; Reproducibility; MR-Linac; Radiotherapy; Functional MRI
MeSH Terms: conditions — Rectal Neoplasms; Pelvic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volunteers (Other): Single arm of volunteers.
  Interventions: Device: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Device: Magnetic Resonance Imaging (MRI) — - Three MRI :
  * two on an MR-Linac 1.5 Tesla (10 to 17 days apart)
  * one on a standard 1.5 Tesla MRI

SUMMARY:
This study evaluates the reliability of functional MRI measurements in pelvic disease through quantifying repeatability and reproducibility, using healthy volunteers. The aim is to provide insights into the consistency of results across sessions and observers, informing the trustworthiness of functional MRI in assessing pelvic disease and particularly rectal cancers and guiding protocol optimization.

DETAILED DESCRIPTION:
Volunteers will be required to complete a questionnaire to ensure their eligibility and safety for undergoing an MRI. This questionnaire, along with safety information, will be reviewed before each MR session.

Subsequently, volunteers will undergo three MRI sessions, ideally two on the same day, with the last session scheduled 10 to 17 days apart from the previous ones. Each session is expected to last approximately 60 minutes (several sequences), and no contrast agent will be injected at any point.

On the first day, volunteers will have an MRI on the 1.5 Tesla MR-Linac Unity (Elekta device) and an MRI on a standard 1.5 Tesla MRI (Siemens). Between days 10 to 17, they will exclusively undergo an MR-Linac session.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 yo
* Healthy
* Volunteer
* Ability to undergo an MRI

Exclusion Criteria:

* < 18yo
* Contraindication to undergoing an MRI (see safety questionnaire)
* Previous pelvic irradiation
* Pelvic pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-13 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Assess the repeatability coefficient (RC) (percentage) | Day 1 and Day 10-17
  Quantitative assessment of the Repeatability Coefficient for functional MRI sequences in rectal tissue, expressed as a percentage.
Assess the reproducibility coefficient (RDC) (percentage) | Day 1 and Day 10-17
  Comparative analysis of Repeatability Coefficient values obtained from distinct MRI devices, providing insights into device-specific variations.

SECONDARY OUTCOMES:
Percentage of variation between the different calculation Methods for Repeatability Coefficient. | Day 1 and Day 10-17
  Comparative evaluation of different calculation methods for the Repeatability Coefficient, highlighting the consistency and discrepancies among methods.
Percentage of variation across various pelvic organs for Repeatability Coefficient. | Day 1 and Day 10-17
  Exploration of Repeatability Coefficients in different pelvic organs, providing insights into the variability of repeatability across distinct anatomical structures.

OTHER OUTCOMES:
Percentage of variation based on sequence types for the Repeatability Coefficients. | Day 1 and Day 10-17
  Comparative assessment of Repeatability Coefficients across different types of functional MRI sequences, elucidating the impact of sequence variations on repeatability.

CONTACTS AND LOCATIONS:
Overall Officials: Madeline A Michel, MD, Principal Investigator — Jules Bordet Institute

IPD SHARING:
Plan to Share IPD: No